CLINICAL TRIAL: NCT02528058
Title: Ultrastructure Analysis of Excised Internal Limiting Membrane in Eyes of Highly Myopia With Myopic Traction Maculopathy
Status: Completed | Type: Observational
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Kyorin Eye Center, Kyorin University
Other Study IDs: Kyorineye018
Record Dates: First submitted 2015-08-16; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Myopic Traction Maculopathy
Keywords: Myopic traction maculopathy
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Excised internal limiting membrane during the surgical treatment for myopic traction maculopathy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Myopic traction maculopathy
  Interventions: Procedure: Vitrectomy with internal limiting membrane peeling

INTERVENTIONS:
Procedure: Vitrectomy with internal limiting membrane peeling

SUMMARY:
The excised ILM from 7 eyes of 7 patients with MTM including 7 eyes with macular retinoschisis and 4 eyes with foveal detachment but without any retinal break underwent vitrectomy with induction of posterior vitreous detachment and ILM peeling was examined to evaluate ultrastructure with electron microscopy.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were patients who underwent vitrectomy and internal limiting membrane peeling for myopic traction maculopathy and had a follow-up for more than 6 months.

Exclusion Criteria:

* The patients with follow-up less than 6 months

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who underwent vitrectomy with internal limiting membrane peeling for myopic traction maculopathy
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2010-06; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Visual acuity before and after surgery | 6 months
  Comparison in logarithm of Minimum Angle of Resolution (logMAR) vision

SECONDARY OUTCOMES:
Retinal reattachment | 6 months
  Resolution of macular retinoschisis and foveal detachment

CONTACTS AND LOCATIONS:
Overall Officials: Akito Hirakata, MD, Principal Investigator — Kyorin Eye Center
Locations (1):
- Makoto Inoue, Mitaka, Tokyo, Japan